CLINICAL TRIAL: NCT03129503
Title: Optical Coherence Tomography in Acute Coronary Syndrome
Acronym: OPTICO-ACS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Berlin Institut of Health (BIH), Germany (Unknown)
Responsible Party: Principal Investigator, David Manuel Leistner, PD Dr. med., Charite University, Berlin, Germany
Other Study IDs: 1.0
Record Dates: First submitted 2017-04-23; First posted 2017-04-26 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Acute Coronary Syndrome; STEMI - ST Elevation Myocardial Infarction; NSTEMI - Non-ST Segment Elevation MI; Atherosclerosis, Coronary
Keywords: Optical coherence tomography (OCT)
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood and coronary thrombus
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute coronary syndrome (ACS): Patients with STE- or NSTE-ACS (acute coronary syndrome)

SUMMARY:
The OPTICO-ACS- study program - combining for the first time in vivo characterization of the ACS-causing "culprit lesion" by intracoronary imaging technique with optical coherence tomography (OCT) and molecular analysis of immune-cells derived from the culprit coronary thrombus and biochemical analyses in patients with acute-coronary-syndrome (ACS).

DETAILED DESCRIPTION:
Using a translational scientific approach the study aims to (a) get a better insight into the different pathophysiological processes in both clinical settings - plaque rupture (RFC) and plaque-erosion (IFC) with focus on to the inflammatory process and molecular mechanisms (b) identify special signatures including clinical and biochemical markers as biomarkers subject to different culprit plaques types and (c) to test its prognostic implications in patients after ACS.

ELIGIBILITY:
Inclusion Criteria:

1. Men and Women (aim: consecutive)
2. Age 18 to 85 years old.
3. ACS as trigger event - (ESC guidelines) being:

   1. Acute cardiac chest pain or angina equivalent consistent with moderate to high-risk unstable angina or myocardial infarction, lasting more than 10 minutes duration during 72 hours before invasive examination AND
   2. Evidence for ACS requiring catheterization documented by a) elevated enzymes (CK-MB or hs-Troponin I/T > 99th percentile or in-/decrease) AND/OR
   3. ECG with ST-depression >1mm in 2 or more contiguous leads after the J-point AND/OR transient ST-elevation >1mm in 2 or more contiguous leads lasting <30 min OR c) STE-ACS with onset < 24 hours previously and chest pain >30 min ST-elevation >1mm in 2 or more contiguous leads or new left bundle block.
4. Written informed consent
5. Patients must have at least coronary one-vessel disease with one angiographically detectable "culprit lesion" (or in case of more > 1 lesion all lesions have to be in one "culprit vessel") in a native coronary vessel requiring PCI. Identification of this lesion as the "culprit lesion" has to be in line with other non-invasive findings (ECG-leads; regional wall motion abnormalities in echocardiography). Other "non-culprit-lesions" are allowed to have significant stenosis requiring interventional revascularization in a staged procedure.

Exclusion Criteria:

1. Active pregnancy.
2. Active sepsis.
3. Acute psychotic disease.
4. Known systolic heart failure with left-ventricular ejection fraction (LV-EF≤ 30 %).
5. Cardiogenic shock or heart failure requiring intubation, inotropes; diuretics or mechanical circulation support.
6. Refractory ventricular arrhythmia requiring pharmacologic or defibrillator therapy.
7. Patients who had received heart transplantation or any other organ transplant or are on waiting list.
8. Renal insufficiency with serum-creatinine ≥ 1.5 mg/dl.
9. Patients with other medical illness (i.e. cancer) or recent history of substance abuse, that may cause non-compliance with the investigational plan, confound the data interpretation or is associated with an anticipated limited life-expectancy less than one year.
10. Prior participation in this study or in other investigational studies, that have not reached its primary endpoint.
11. Unprotected left main- CAD with ≥ 50% stenosis.
12. ACS with culprit lesion in a bypass graft or ACS caused by stent-thrombosis.
13. Extent and severity of CAD is such that investigator believes it is likely that bypass surgery will be required within 1 year of enrollment.
14. No suitable anatomy of "culprit lesion" for OCT:

    * severe calcification or extreme tortuosity of "culprit lesion".
    * culprit lesion with very distal location.
    * infarct vessels with an diameter > 4 mm or < 2 mm.
    * STE-ACS: "No-reflow" (TIMI 0-I) after thrombus aspiration/slight pre- dilatation

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: ACS Patients at Charité University Hospital including all sites
  * Campus Benjamin Franklin (CBF)
  * Campus Virchow Klinikum (CVK)
  * Campus Mitte (CCM)
Sampling Method: Non-Probability Sample
Enrollment: 414 (Estimated)
Dates: Start 2017-04-28 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular Events (MACCE) | 2 years after ACS
  powered

SECONDARY OUTCOMES:
Rehospitalization Rate for Angina pectoris | 2 years after ACS
Major adverse cardiovascular Events (MACCE) | 30 days, 90 days, 12 months and 5 years after ACS
Intima /media thickness | Day 90 after ACS
  by sonography
Global and regional left-ventricular systolic and diastolic function | After ACS and 90 days after ACS
  by echocardiography
Frequency and severity of angina | at day 90,12 and 24 months after ACS
  by Seattle Angina questionnaire
Pulse-wave-velocity (PWV), Augmentation index (AI) and Sub-endocardial Viability Ratio (SEVR). | Day 90 after ACS
  by SphygmoCor system
Lesion Coverage | within 6 weeks to 3 months
  by OCT

CONTACTS AND LOCATIONS:
Overall Officials: David M Leistner, MD, Study Chair — Charite - University Medicine Berlin - Department for cardiology; Ulf Landmesser, MD, Study Chair — Charite - University Medicine Berlin - Department for cardiology
Locations (3):
- Germany (3):
  - Charite University Campus Mitte, Berlin
  - Charite University Campus Benjamin Franklin, Berlin
  - Charite University Campus Virchow-Klinikum, Berlin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seppelt C, Abdelwahed YS, Meteva D, Nelles G, Stahli BE, Erbay A, Krankel N, Sieronski L, Skurk C, Haghikia A, Sinning D, Dreger H, Knebel F, Trippel TD, Krisper M, Gerhardt T, Rai H, Klotsche J, Joner M, Landmesser U, Leistner DM. Coronary microevaginations characterize culprit plaques and their inflammatory microenvironment in a subtype of acute coronary syndrome with intact fibrous cap: results from the prospective translational OPTICO-ACS study. Eur Heart J Cardiovasc Imaging. 2024 Jan 29;25(2):175-184. doi: 10.1093/ehjci/jead154. PMID 37395586
- [Derived] Leistner DM, Krankel N, Meteva D, Abdelwahed YS, Seppelt C, Stahli BE, Rai H, Skurk C, Lauten A, Mochmann HC, Frohlich G, Rauch-Krohnert U, Flores E, Riedel M, Sieronski L, Kia S, Strassler E, Haghikia A, Dirks F, Steiner JK, Mueller DN, Volk HD, Klotsche J, Joner M, Libby P, Landmesser U. Differential immunological signature at the culprit site distinguishes acute coronary syndrome with intact from acute coronary syndrome with ruptured fibrous cap: results from the prospective translational OPTICO-ACS study. Eur Heart J. 2020 Oct 1;41(37):3549-3560. doi: 10.1093/eurheartj/ehaa703. PMID 33080003